CLINICAL TRIAL: NCT03820024
Title: The MOVES Trial: MOtiVating Endometrial Cancer Survivors With Activity Monitors and Tailored Feedback
Brief Title: MOtiVating Endometrial Cancer Survivors With Activity Monitors and Tailored Feedback
Acronym: MOVES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LCCC 1614
Record Dates: First submitted 2018-10-16; First posted 2019-01-29 (Actual); Results first posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored Feedback Messages (Experimental): Participants randomized to the message arm will begin receiving encouragement and reminder UNC CHART messages to increase physical activity weekly based on the CHART algorithm (Appendix 1). Participants on the feedback arm will receive 1 message per week during the 3-month study period.
  Interventions: Behavioral: Tailored Feedback Messages
- No Messages (No Intervention): No feedback messages

INTERVENTIONS:
Behavioral: Tailored Feedback Messages — Participants randomized to the message arm will begin receiving encouragement and reminder UNC CHART messages to increase physical activity weekly. Participants on the feedback arm will receive 1 message per week during the 3-month study period.
  Arms: Tailored Feedback Messages

SUMMARY:
Overweight and obese endometrial cancer (EC) survivors at the University of North Carolina (UNC) at Chapel Hill will be approached for tailored feedback fitness intervention. The investigators plan to enroll 36 women (18 in each arm) to evaluate if receipt of weekly tailored feedback messages can improve physical activity in EC survivors. It is hypothesized that women receiving the feedback message intervention will increase step counts from baseline more than 2,000 steps compared to women in the non-intervention arm.

DETAILED DESCRIPTION:
Objectives:

* To assess if a tailored feedback fitness intervention can increase physical activity in EC survivors from baseline to 12 weeks post-baseline
* To determine the acceptability of the fitness intervention in EC survivors through a completion survey.
* To assess if a tailored feedback message fitness intervention can (1) decrease BMI, (2) reduce waitst to hip (W.H) ratios, (3) improve quality of life (QOL) and (4) improve serum metabolic markers (insulin, glucose and low density lipoprotein (LDL) in EC survivors.

ELIGIBILITY:
Inclusion Criteria:

* Be over the age of 18 years
* Have a confirmed diagnosis of endometrial cancer and have completed therapy (surgery, chemotherapy or radiation) within the past 6 months
* Have no current evidence of endometrial cancer
* Have a BMI 25 kg/m2 or greater
* Have approval from their treating physician to engage in moderate-intensity physical activity.
* Have a smart phone with Bluetooth capabilities turned on
* Have access to email

Exclusion Criteria:

* Are currently undergoing treatment for their cancer
* Are unable to read a sample message aloud
* Do not have a computer or smart phone with Bluetooth capabilities
* Are pregnant
* Have a history of angina or palpitations with exertion
* Have a history of uncontrolled pulmonary disease (COPD or asthma)
* Have one or more significant medical conditions that in the physician's judgment preclude participation in the walking intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2020-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Clark, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- North Carolina Cancer Hospital, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 9/28/2018 to 12/23/2019
Pre-assignment Details: Thirty-nine participants were consented
Period: Overall Study
Arm/Group | Tailored Feedback Messages | No Messages
Started | 19 | 20
Completed | 18 | 18
Not Completed | 1 | 2
Not completed — Physician Decision | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tailored Feedback Messages | No Messages | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Full Range); unit: years] | 55.3 [36 to 76] | 56.4 [43 to 68] | 55.7 [36 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 12 | 13 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Change in Steps in Endometrial Cancer Survivors During 12 Week Intervention
Description: Steps recorded on a fitness tracker at week 1 and week 13
Time Frame: 13 weeks
Measure: Mean (Standard Error); unit: Change in steps
Arm/Group | Tailored Feedback Messages | No Messages
Number analyzed (Participants) | 18 | 18
Change in steps | 1037 (0.02) | 309 (0.4)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Tailored Feedback Messages | No Messages
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-13): https://cdn.clinicaltrials.gov/large-docs/24/NCT03820024/Prot_SAP_000.pdf